CLINICAL TRIAL: NCT00969969
Title: A Study to Evaluate the Effectiveness and Safety of an Implant in the Treatment of Osteoarthritis of the Great Toe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cartiva, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTC-0031
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Osteoarthritis of First Metatarsalphalangeal Joint
Keywords: First MTP Joint; Hallux Rigidus; Hallux Limitus; Cartilage Replacement; Osteoarthritis; First MTP Joint Osteoarthritis; Big Toe Pain
MeSH Terms: conditions — Hallux Rigidus; Hallux Limitus; Osteoarthritis | interventions — Arthrodesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arthrodesis (Active Comparator): Fusion
  Interventions: Device: Arthrodesis
- Cartiva (Experimental): Synthetic Cartilage Implant
  Interventions: Device: Cartiva

INTERVENTIONS:
Device: Arthrodesis — arthrodesis using screws and/or a plate
  Arms: Arthrodesis
Device: Cartiva — Cartiva Synthetic Cartilage Implant
  Arms: Cartiva

SUMMARY:
This study will evaluate whether Cartiva is an effective treatment for individuals with osteoarthritis of the great toe.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Osteoarthritis of the first metatarsophalangeal joint and is a candidate for arthrodesis
* Presence of good bone stock
* Capable of completing self-administered questionnaires

Exclusion Criteria:

* < 18 years of age
* Osteoarthritis of the first metatarsophalangeal joint, though is not a candidate for arthrodesis
* Active bacterial infection of the foot
* Additional ipsilateral limb (hip, knee, ankle, or foot) pathology that requires active treatment (surgery or brace)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2009-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
VAS, FAAM, Safety | up to 2 years
  The individual components of the primary outcome measures will be Visual Analog Scale (VAS) Pain, Foot and Ankle Ability Measure (FAAM) Sports sub-scale score and absence of key safety issues.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Baumhauer, Principal Investigator — University of Rochester
Locations (12):
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Horizon Health Network, Fredericton, New Brunswick
  - Queen Elizabeth Science Centre, Halifax, Nova Scotia
  - St. Michael's Hospital, Toronto, Ontario
- United Kingdom (6):
  - Frimley Park Hospital - Surrey Foot and Ankle Clinic, Frimley, Camberley
  - St. George's Hospital, Tooting, London
  - Royal National Orthopaedic Hospital - Stanmore Foot & Ankle Clinic, Stanmore, Middlesex
  - Northern General Hospital NHS Trusts - Sheffield Orthopaedics, Sheffield, South Yorkshire
  - Royal Surrey County Hospital, Guildford, Surrey
  - Torbay Hospital, South Devon, Torquay

IPD SHARING:
Plan to Share IPD: No